CLINICAL TRIAL: NCT04897646
Title: Evaluation of a CPAP Telemonitoring Algorithm for Newly Treated Patients: the TELEAP1 Multicenter Cohort Pilot Study
Brief Title: The TELEAP1 CPAP-telemonitoring Study
Acronym: TELEAP1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: ADENE, Montpellier (Unknown); AGIR à dom, Meylan (Unknown); ASTEN sante, Pays de la Loire (Unknown); ELIA medical, Cesson-Sévigné (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0082
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep apnea; Continuous Positive Airway Pressure,; Telemedicine; COVID 19; observance; leaks; apnea hypopnea index.
MeSH Terms: conditions — Sleep Apnea, Obstructive; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: SFRMS/SPLF CPAP-telemonitoring diagnosis/therapeutic algorithm. — In 2020, a working group from the Société Française de Recherche et de Médecine du Sommeil (SFRMS) and the Société de Pneumologie de Langue Française (SPLF) have proposed a CPAP-telemonitoring diagnosis/therapeutic algorithm for newly treated patients with obstructive sleep apnea.
  The algorithm is exhasutively described in the following published article: Prigent, A., Gentina, T., Launois, S., et al. [Telemonitoring in continuous positive airway pressure-treated patients with obstructive sleep apnoea syndrome: An algorithm proposal]. Rev. Mal. Respir., 2020, 37: 550-560.

SUMMARY:
TELEAP1 is a multicenter cohort pilot-study designed to evaluate the impact of a published SFRMS/SPLF CPAP-telemonitoring diagnosis/therapeutic algorithm on the CPAP-compliance of newly treated patients with obstructive sleep apnea..

DETAILED DESCRIPTION:
Continuous Positive Airway Pressure (CPAP)-devices can track compliance, but also leaks and residual Apnea-Hypopnea-Index (AHIflow) values. CPAP tracking systems seem intuitively useful, but there are few data demonstrating the benefit of such systems in improving CPAP-compliance and/or patients quality of life.

In 2020, a working group from the Société Française de Recherche et de Médecine du Sommeil (SFRMS) and the Société de Pneumologie de Langue Française (SPLF) have proposed a CPAP-telemonitoring diagnosis/therapeutic algorithm for newly treated patients with obstructive sleep apnea.

In order to describe and evaluate the impact of this SFRMS/SPLF-algorithm (not only on the patient but also on the home care provider activity), a one year multicenter cohort pilot-study (TELAP1-study) was set up.

ELIGIBILITY:
Inclusion criteria:

* 18 years of age or older
* Patient newly CPAP-treated and eligible for care and for the reimbursement by the French Social Security rules
* Signed informed consent

Exclusion criteria:

* Previous CPAP-treatment
* Pregnancy
* Inability to understand the nature and aims of the study or to communicate with the investigator
* Simultaneous participation in another trial with an exclusion clause to participate in another trial
* No affiliation with the French social security regime
* Loss of personal capacity resulting in state protection
* Deprivation of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the study are newly CPAP-treated with a diagnosis of obstructive sleep apnea.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
CPAP-complianceversus corresponding 2019 weeks (h/days) | 4 months
  CPAP-compliance (hour/day) reported by the CPAP-software for the last 28 days

SECONDARY OUTCOMES:
AHIflow | 4 months
  AHIflow (events/hour) reported by the CPAP-software for the last 28 days
CPAP-adherence | 12 months
  CPAP-adherence defined as the % of patients with a CPAP-adherence >4h/day, CPAP-adherence reported by the CPAP-software for the last 28 days.
CPAP-leaks | 4 months
  important leaks (l/min or % or min/days) reported by the CPAP-software for the last 28 days
CPAP-leaks | 12 months
  important leaks (l/min or % or min/days) reported by the CPAP-software for the last 28 days
Patient subjective sleepiness | 4 months
  reported by the patient using the Epworth Sleepiness Scale (0-24)
Patient subjective sleepiness | 12 months
  reported by the patient using the Epworth Sleepiness Scale (0-24)
Patient subjective depression | 12 months
  reported by the patient using the Pichot Depression Scale (0-13)
Patient subjective insomnia | 4 months
  reported by the patient using the Insomnia Severity Scale (0-28)
Patient subjective insomnia | 12 months
  reported by the patient using the Insomnia Severity Scale (0-28)
CPAP-compliance | 12 months
  CPAP-compliance (hour/day) reported by the CPAP-software for the last 28 days
Unplanned patient phone call | Day 0 to 360
  unplanned patient phone call with the technician regardless of the reason
Unplanned technician phone call | Day 0 to 360
  unplanned technician phone call with the patient regardless of the reason
Unplanned patient visit | Day 0 to 360
  unplanned patient visit to the care provider regardless of the reason
Unplanned technician visit | Day 0 to 360
  unplanned technician visit to the patient regardless of the reason
CPAP telemonitoring alarm | Day 0 to 360
  number and type (cpap observance < 4h for the last 7 days, and or IAHflow >10/h for the last 7 days, and or important leaks for the last 7 days)
Interface-type change | Day 0 to 360
  description of the interface-type change (nasal, nasal pillows, oronasal) regardless of the reason
Pressure settings modification | Day 0 to 360
  Change in the CPAP-pressure settings regardless of the reason
CPAP-mode modification | Day 0 to 360
  Change in the CPAP mode (constant or auto-CPAP) regardless of the reason

CONTACTS AND LOCATIONS:
Overall Officials: Dany Jaffuel, MD,PhD, Principal Investigator — Montpellier University Hospitals; Fréderic Gagnadoux, Study Director — University Hospital, Angers; Arnaud Prigent, Principal Investigator — Polyclinique Saint Laurent - Rennes; Renaud Tamisier, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No